CLINICAL TRIAL: NCT01625923
Title: A Pilot Study on the Efficacy and Safety of Olanzapine in Improving Symptoms and Gastric Motility in Gastroparesis
Brief Title: A Pilot Study on the Efficacy and Safety of Olanzapine in Gastroparesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment numbers
Sponsor: University of Michigan (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Allen Lee, Clinical Lecturer, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACG-SP-002-2012
Record Dates: First submitted 2012-06-18; First posted 2012-06-22 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Idiopathic Gastroparesis
Keywords: Gastroparesis; Idiopathic; Olanzapine
MeSH Terms: conditions — Gastroparesis | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olanzapine (Experimental): An open-label pilot study of 20 consecutive subjects ages 18 - 70 with documented delayed gastric emptying within the past 2 years and history of nausea, vomiting, bloating, anorexia, early satiation, post-prandial fullness, and weight loss for at least 6 months without structural or organic cause will be enrolled.
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Subjects will initially start on olanzapine 2.5 mg per mouth daily. Subjects will return on days 7 and 14 to determine response to medication and medication dose can be increased to 5 mg and 10 mg, respectively, based on incomplete symptom response (mean change GCSI-DD < 0.5). The total dose of olanzapine will not exceed 10 mg daily during this study and subjects will continue on treatment for a total of 8 weeks.
  Other Names: Zyprexa

SUMMARY:
Gastroparesis is a disorder characterized by impaired gastric emptying in the absence of obstruction in the proximal GI tract. It is a common condition affecting up to 5 million persons in the United States alone. Despite this, metoclopramide is currently the only FDA approved medication for the treatment of gastroparesis. However, the evidence supporting metoclopramide in gastroparesis is fairly weak and was recently issued a black box warning because of potential irreversible side effects. There is clearly an urgent need for newer therapeutic options with better efficacy and tolerability. Olanzapine is a second generation anti-psychotic that is currently FDA approved for the treatment of schizophrenia and bipolar disorder. Because of actions at several receptors throughout the body, including dopamine and serotonin receptors, Olanzapine may provide anti-nausea and pro-motility effects in the stomach. Long-term use of olanzapine may also increase plasma levels of ghrelin. Ghrelin is a hormone produced by the gut that stimulates appetite and has also been shown to have beneficial effects on gastroparesis. The investigators hypothesize that olanzapine will be effective and safe in controlling symptoms as well as stimulate appetite and weight gain in gastroparesis. The investigators also hypothesize that olanzapine will stimulate gastric motility. Finally, the investigators hypothesize that olanzapine will modulate the secretion of ghrelin in gastroparesis. This pilot study may provide further information on the efficacy and safety of olanzapine in gastroparesis which could be utilized in a larger randomized, prospective study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 70 years of age
* Must have a > or = 6 month history of relevant symptoms of gastroparesis, (e.g., chronic post-prandial fullness, early satiety, postprandial nausea), patients will have a mean of the daily scores over a minimum of 7 days indicating > or = mild (2) and < or = severe (4) post-prandial fullness assessed using the GCSI-DD during the screening period prior to randomization
* Documented abnormal gastric emptying within the past 2 years
* Has gastroparesis at screening (gastric half-time of emptying > upper limit of normal as determined by wireless motility capsule)
* BMI between 18 - 30 kg/m2
* A female subject is eligible to participate if she is of non-childbearing potential or child-bearing potential and agrees to use one of the approved contraception methods. Female patients must agree to use contraception for at least 5 days following the last dose of study medication
* Subject has never had a gastrectomy, nor major gastric surgical procedure or any evidence of bowel obstruction or strictures within the previous 12 months
* Dosage of any concomitant medications has been stable for at least 3 weeks.
* Estimated (or measured) glomerular filtration rate ≥ 30 mL/min
* QTcB or QTcF < 450 msec or QTc < 480 msec in patients with Bundle Branch. Block based on single or average QTc value of triplicate values obtained over a brief recording period
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN; normal CBC, TSH, and prolactin levels

Exclusion Criteria:

* History of diabetes mellitus or hyperglycemia
* History of cardiovascular or cerebrovascular disease
* History of hyperlipidemia
* History of cardiac arrhythmia or long QT syndrome
* History of seizure disorder
* History of hyperprolactinemia
* History of renal dysfunction
* History of hepatic impairment
* History of schizophrenia, bipolar disorder, or previous use of olanzapine
* History of Parkinson's disease, dementia or severe cognitive impairment
* History of GI surgery or placement of gastric pacemaker
* History of cardiac pacemaker or implantable cardiac defibrillator
* History of eating disorder
* History of intrapyloric botulinum toxin injections
* Subject is on chronic enteral or parenteral feeding
* Subject has pronounced dehydration
* Subject has evidence of severe cardiovascular autonomic neuropathy (e.g. history of recurrent syncope in the last 6 months)
* Use of medications potentially influencing upper gastrointestinal motility or appetite within one week of the study (e.g., prokinetic drugs, macrolide antibiotics (erythromycin), GLP-1 mimetics)
* Regular opiate use
* Subjects who are taking drugs that potentially interact with olanzapine including diazepam, lorazepam, alcohol, carbamazepine, fluvoxamine, olanzapine and fluoxetine in combination, CNS acting drugs, levodopa and dopamine agonist, and olanzapine when used in combination with lithium or valproate
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease or other condition that would in the opinion of the investigator or medical monitor make the subject unsuitable for inclusion in this clinical study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator would make the subject unsuitable for inclusion in this clinical study
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day time-period
* Pregnant females as determined by positive serum or urine hCG test (from the first urine of the day) at screening or prior to dosing
* Lactating females
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subject is unable to swallow pills

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Lee, MD, Principal Investigator — University of Michigan; Braden Kuo, MD, Principal Investigator — Massachusetts General Hospital; William Hasler, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine: Subjects were enrolled to receive olanzapine open-label for 8 weeks. Subjects were initially started on olanzapine 2.5 mg by mouth daily at bedtime. Subjects returned on days 7 and 14 to determine response to medication. Medication dose was increased to 5 mg on day 7 and 10 mg on day 14, respectively, if there was incomplete symptom response, which was defined as a mean change in GCSI-DD score < 0.5 from baseline.
Period: Overall Study
Arm/Group | Olanzapine
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Olanzapine: Olanzapine
Arm/Group | Olanzapine
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 40.3 [26 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean BMI
Description: Subjects will undergo regular testing of blood glucose, insulin, hemoglobin (Hgb) A1c, body mass index (BMI), liver enzymes, thyroid stimulating hormone (TSH), and prolactin levels during the study as well as after treatment completion to determine the safety of the medication. All adverse events will be compiled to investigate the tolerability of the medication.
Time Frame: 8 weeks
Population: Change in mean BMI
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Olanzapine
Number analyzed (Participants) | 3
kg/m^2
  Baseline BMI | 23.5 (3.4)
  BMI at Week 8 | 24.9 (3.6)

2. Primary Outcome: Mean GCSI-DD Before/After Treatment With Olanzapine
Description: The investigators will utilize the gastroparesis cardinal symptom index daily diary (GCSI-DD) to compare severity of symptoms before and after treatment with olanzapine. The total GCSI-DD is a validated questionnaire that measures the daily relevant symptoms of gastroparesis and ranges from 0 (no symptoms) to 5 (severe symptoms).
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Olanzapine
Number analyzed (Participants) | 3
score on a scale
  Baseline GCSI-DD Score | 3.11 (0.42)
  GCSI-DD Score After Intervention | 2.17 (0.17)
Statistical Analysis 1: Comparison: Olanzapine; Test type: Other — T-test comparing GCSI-DD scores before/after intervention; p = .06, t-test, 2 sided

3. Primary Outcome: Change in Mean Serum Glucose
Description: as for outcome 1
Time Frame: 8 weeks
Population: Change in mean serum glucose
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Olanzapine
Number analyzed (Participants) | 3
mg/dl
  Baseline Serum Glucose | 90.5 (0.7)
  Serum Glucose at Week 8 | 90.5 (0.7)

4. Secondary Outcome: Change in Mean Gastric Emptying Time
Description: The investigators aim to test gastric motility, including gastric emptying and antroduodenal contractility parameters, by wireless motility capsule (WMC) before and at the completion of the study to determine if olanzapine has any pro-motility effects in gastroparesis.
Time Frame: 8 weeks
Population: Change in mean gastric emptying time by WMC
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Olanzapine
Number analyzed (Participants) | 3
minutes
  Baseline GET (minutes) | 468.3 (233.4)
  GET at Week 8 (minutes) | 563.3 (582.6)

5. Secondary Outcome: Change in Mean Ghrelin Levels Over Time
Description: The investigators seek to determine whether olanzapine promotes secretion of ghrelin in gastroparesis.
Time Frame: 8 weeks
Population: Change in mean ghrelin levels over time
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Olanzapine
Number analyzed (Participants) | 3
pg/ml
  Baseline plasma ghrelin (pg/ml) | 615.7 (339.1)
  Plasma ghrelin at week 8 (pg/ml) | 577.0 (253.4)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Olanzapine
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olanzapine (N=3)
Fatigue (General disorders) | 2
Weight gain (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT01625923/Prot_SAP_000.pdf